CLINICAL TRIAL: NCT05108766
Title: A Phase Ⅲ, Multicenter, Randomized, Double-blind, Placebo Controlled Trial Evaluating the Efficacy and Safety of Tildrakizumab in the Treatment of Chinese Subjects With Moderate to Severe Plaquetype Psoriasis
Brief Title: A Phase Ⅲ Study to Evaluate Tildrakizumab in the Treatment of Chinese Subjects With Moderate to Severe Plaquetype Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen Kangzhe Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tildra-PsO-001
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — tildrakizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tildrakizumab (Experimental): Subjects will receive 100 mg subcutaneous (SC) Tildrakizumab at Week 0 and Week 4, 100 mg subcutaneous placebo at Week 12. Subjects entered the extension study after completion of the base study and will receive 100 mg subcutaneous Tildrakizumab at Week 16, 28, 40, and 52.
  Interventions: Drug: Tildrakizumab 100 mg
- Placebo (Placebo Comparator): Subjects will receive 100 mg subcutaneous placebo at Week 0 and Week 4, and 100 mg subcutaneous Tildrakizumab at Week 12. Subjects entered the extension study after completion of the base study and will receive 100 mg subcutaneous Tildrakizumab at Week 16, 28, 40, and 52.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tildrakizumab 100 mg — Tildrakizumab 100 mg administered SC. Each PFS contains 1 mL of solution, tildrakizumab 100 mg/mL.
  Other Names: SCH 90022; MK-3222
  Arms: Tildrakizumab
Drug: Placebo — Matching placebo to tildrakizumab administered SC
  Arms: Placebo

SUMMARY:
This is a phase Ⅲ, randomized, double-blind, placebo-controlled, parallel design, multicenter trial to evaluate the efficacy, safety, tolerability, and immunogenicity of subcutaneous Tildrakizumab in subjects with moderate to severe chronic plaque psoriasis.

The trial was divided into two parts: the base study (Week 0- Week 12) and the extension study (Week 13- Week 54).

DETAILED DESCRIPTION:
Base Study： 220 subjects were randomized in a 1: 1 ratio into the trial, and the treatment group received 100 mg subcutaneous Tildrakizumab at Week 0 and Week 4, 100 mg subcutaneous placebo at Week 12, while the placebo group received 100 mg subcutaneous placebo at Week 0 and Week 4, and 100 mg subcutaneous Tildrakizumab at Week 12, and subjects will be evaluated for efficacy, safety, tolerability, and immunogenicity as specified in this protocol. At the end of the base study, procedures such as data cleaning, locking and unblinding of base study data were performed.

Extension Study： Subjects entered the extension study after completion of the base study and will receive 100 mg subcutaneous Tildrakizumab at Week 16, 28, 40, and 52, and will be evaluated for efficacy, safety, tolerability, and immunogenicity by the investigator according to the regulations of this study.

At the end of the extension study, all data from the extension study will be entered into the database, after the data is reviewed, cleaned, and locked, the entire trial will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must give a written, signed and dated informed consent.
2. Subject must be 18-70 years of age, of either sex.
3. Diagnosis of predominantly plaque psoriasis for over 6 months (Plaque psoriasis in stable phase, and in non-progressive phase as determined by subject interview and confirmation of diagnosis through physical examination by investigator).
4. Subject is considered to be a candidate for phototherapy or systemic therapy.
5. Psoriasis BSA involvement ≥ 10% at baseline.
6. PASI score ≥ 12 at baseline.
7. PGA of at least moderate disease (≥ 3) at baseline.
8. No history of active TB or symptoms of TB; No recent history of intimate contact with patients with active TB;
9. Subject is a male or a non-sterilized, pre-menopausal female and agrees to abstain from heterosexual activity OR use a medically accepted method of contraception OR use appropriate effective contraception as per local regulations or guidelines. Medically accepted methods of contraception include, but are not limited to, condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed IUD, inert or copper-containing IUD, hormone-releasing IUD, systemic hormonal contraceptive, and surgical sterilization (e.g., hysterectomy or tubal ligation).
10. For a woman of childbearing potential, a negative serum pregnancy test at Screening/baseline.

Exclusion Criteria:

1. Presence of predominantly non-plaque forms of psoriasis：guttate psoriasis, erythrodermic psoriasis, pustular psoriasis, medication-induced or medication-exacerbated psoriasis.
2. Subjects who are expected to require additional topical therapy, phototherapy, or systemic therapy other than trial drug for the treatment of psoriasis during the trial.
3. Presence of any infection or history of recurrent infection requiring treatment with systemic antibiotics within 2 weeks prior to Screening, or severe infection (e.g., pneumonia, cellulitis, bone, or joint infections) requiring hospitalization or treatment with IV antibiotics within 8 weeks prior to Screening.
4. Subject is known to be allergic to Tildrakizumab or related excipients.
5. Women of childbearing potential who are pregnant or are lactating, female subject or male subject with partner intend to become pregnant (during the trial OR within 6 months of the last administration of the trial drug).
6. Positive human immunodeficiency virus (HIV) antibody (HIV Ab)test result and/or positive Treponema pallidum-specific antibody test result, and/or positive hepatitis C virus antibody (HCV Ab) test result with positive HCV-RNA reverse transcription polymerase chain reaction test result, indicating a past or current infection of hepatitis C virus; and/or positive result of hepatitis B surface antigen (HbsAg) , or positive result of hepatitis B core antibody (HBcAb) with positive result of HBV-DNA polymerase chain reaction test, indicating an current infection of HBV; .
7. Subject has the following clinically significant abnormal laboratory tests according to the investigators' evaluation.
8. Prior malignancy or concurrent malignancy (excluding successfully treated basal cell carcinoma, squamous cell carcinoma of the skin in situ, squamous cell carcinoma with no evidence of recurrence within 5 years or carcinoma in situ of the cervix that has been adequately treated).
9. Subject who has received a live attenuated vaccine within 4 weeks prior to first dose or who intends to receive live attenuated vaccine during the trial.
10. Subject who is currently participating in another interventional clinical trial or has participated in an interventional clinical trial within 4 weeks prior to first dose.
11. The subject is among the personnel of the investigational site or sponsor/designee directly involved with this trial.
12. Within 6 months prior to Screening, subject has any significant organ dysfunction or clinically significant laboratory abnormalities that place the subject at unacceptable risk for participation in a trial of an immunomodulatory therapy in the judgment of the investigator.
13. Within 6 months prior to screening, subject has decompensated cardiac insufficiency (New York Heart Association (NYHA) class III or IV) ; presence of unstable angina, myocardial infarction, history of coronary artery bypass graft, or coronary stent implantation; presence of cardiac arrhythmias (such as long QT syndrome, etc.) that requires medical treatment and is evaluated as ineligible for participation in this clinical trial according to the investigator; hospitalization due to an acute cardiovascular event, cardiovascular illness, or cardiovascular surgery.
14. Subject has sustained uncontrolled hypertension (systolic blood pressure of ≥ 160 mm Hg and/or diastolic blood pressure of ≥ 100 mm Hg at screening) and/or uncontrolled diabetes (fasting glucose ≥ 7 mmol/L and HbA1C ≥ 7.0%).
15. Subject who, has history of alcohol abuse (i.e., alcohol abuse > 2 units of alcohol per day (1 unit = 360 mL of beer or 45 mL of alcohol in 40% of Chinese spirits or 150 mL of wine)) or history of drug abuse.
16. Subject was treated with IL-23/Th-17 pathway inhibitors, including p40, p19 and IL-17 antagonists and failed.
17. Subject has current signs or symptoms of severe, progressive, or uncontrollable renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic and cerebral and/or psychiatric illness.
18. Subject is in other conditions deemed unsuitable for the trial by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with at least 75% improvement in the Psoriasis Area and Severity Index (PASI 75) at Week 12 from baseline in each group. | Week 12
  The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status.

SECONDARY OUTCOMES:
The proportion of subjects in each group with a Physician's Global Assessment (PGA) score of "clear" or "minimal" and at least a 2-grade reduction from baseline at Week 4, 8, and 12. | Week 4, 8, and 12
  The PGA is used to determine the overall severity of a participant's psoriasis lesions at a given time point. Overall lesions will be graded for thickness, erythema, and scaling on a scale from 0 to 5. The sum of the 3 scales will be divided by 3 to obtain the PGA score. PGA is assessed as: 0= Cleared, except for residual discoloration. 1= Minimal, majority of lesions have individual scores that average 1. 2 =Mild, majority of lesions have individual scores that average 2. 3= Moderate, majority of lesions have individual scores that average 3. 4= Marked, majority of lesions have individual scores that average 4. 5= Severe, majority of lesions have individual scores that average 5.
Change from baseline in the Dermatology Life Quality Index (DLQI) at Week 12 in each group. | Week 12
  The DLQI questionnaire consists of 10 questions, where each question is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life.
Change from baseline in PASI 75, 90, and 100 responses over time from Week 0 to Week 12 in each group. | Week 12
  The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status.

OTHER OUTCOMES:
Work Productivity Loss Questionnaire (WPLQ) at Week 12, 28, 40, 52 in each group. | Week 12, 28, 40, 52
  The WPLQ provided information for evaluation of the impact of the subject's psoriasis on their work.
Mean variations and change from baseline in PASI score over time from Week 0 to Week 52 in each group. | Week 0 to Week 52
  The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status.
Change from baseline in the proportion of subjects with a PGA score of "clear" or "minimal" and at least a 2-grade reduction from baseline at weeks 28, 40 and 52 in each group. | Week 28, 40, 52
  The PGA is used to determine the overall severity of a participant's psoriasis lesions at a given time point. Overall lesions will be graded for thickness, erythema, and scaling on a scale from 0 to 5. The sum of the 3 scales will be divided by 3 to obtain the PGA score. PGA is assessed as: 0= Cleared, except for residual discoloration. 1= Minimal, majority of lesions have individual scores that average 1. 2 =Mild, majority of lesions have individual scores that average 2. 3= Moderate, majority of lesions have individual scores that average 3. 4= Marked, majority of lesions have individual scores that average 4. 5= Severe, majority of lesions have individual scores that average 5.
Change from baseline in DLQI at Week 28, 40, 52 in each group. | Week 28, 40, 52
  The DLQI questionnaire consists of 10 questions, where each question is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life.
Change from baseline in PASI 75, 90, 100 response at Week 28, 40, 52 in each group. | Week 28, 40, 52
  The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the area of involvement. Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status.
The positive rate and change of anti-drug antibodies in subjects treated with Tildrakizumab at Week 0, 4, 12, 28, 40 and 52 in each group. | Week 0, 4, 12, 28, 40 and 52
  Observe and evaluate the positive rate and change of anti-drug antibodies of Tildrakizumab in patients after treatment.
  Blood sampling point design: Anti-drug antibodies:
  Blood samples will be collected on Day 1 of Week 0, Day 1 (± 3 days) of Week 4 and Week 12, Day 1 (± 5 days) of Week 28, and Day 1 (± 7 days) of Week 40 and Week 52 prior to dosing or at the Early Withdrawal Visit, with 5 mL of whole blood collected each, divided into two tubes (test tube and backup tube) after centrifugation.
The positive rate and change of neutralizing antibodies in subjects treated with Tildrakizumab at Week 0, 4, 12, 28, 40 and 52 in each group. | Week 0, 4, 12, 28, 40 and 52
  Observe and evaluate the positive rate and change of neutralizing antibodies of Tildrakizumab in patients after treatment.
  Blood sampling point design: neutralising antibodies (neutralising antibodies should be tested if anti-drug antibodies are positive):
  Blood samples will be collected on Day 1 of Week 0, Day 1 (± 3 days) of Week 4 and Week 12, Day 1 (± 5 days) of Week 28, and Day 1 (± 7 days) of Week 40 and Week 52 prior to dosing or at the Early Withdrawal Visit, with 5 mL of whole blood collected each, divided into two tubes (test tube and backup tube) after centrifugation.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Air Force Medical University of PLA, Xi'an, China

REFERENCES:
- [Derived] Yu C, Geng S, Yang B, Deng Y, Li F, Kang X, Bi M, Zhang F, Zhao Y, Pan W, Tian Z, Xu J, Zhang Z, Yu N, Duan X, Guo S, Sun Q, Li W, Tao J, Liu Z, Yin Y, Wang G. Tildrakizumab for moderate-to-severe plaque psoriasis in Chinese patients: A 12-week randomized placebo-controlled phase III trial with long-term extension. Chin Med J (Engl). 2024 May 20;137(10):1190-1198. doi: 10.1097/CM9.0000000000002873. Epub 2024 Jan 9. PMID 38192233